CLINICAL TRIAL: NCT06337591
Title: Diagnostic Performance of the Vesical Imaging-Reporting and Data System (VI-RADS) in Detecting Muscle-invasive Bladder Tumour (MIBC) in Clinical Practice: Comparison With Transurethral Resection of Bladder Cancer (TURB) and Evaluation of Diagnostic Accuracy According to Tumour Location
Acronym: VI-RADS
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_003_2024
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; TURB; VI-RADS
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with suspected primary bladder tumour (TV) at cystoscopy
  Interventions: Procedure: VI-RADS

INTERVENTIONS:
Procedure: VI-RADS — Patients with suspected bladder cancer underwent multiparametric magnetic resonance imaging (mMRI) and vescical imaging reporting and data system (VI-RADS) score calculation. After trans-urethral resection of bladder (TURB), the results of biopsy were compared to the VI-RADS score to verify their concordance.

SUMMARY:
VI-RADS was an observational, prospective, multicenter, no profit study. The aim of the study was to clarify the clinical validity of the Vesical Imaging-Reporting and Data System (VI-RADS) for the assessment of muscle invasion (MI) status in comparison with transurethral resection of bladder cancer (TURB) and to evaluate the diagnostic accuracy of the score according to the specific tumour location.

DETAILED DESCRIPTION:
The VI-RADS (bladder imaging-reporting and data system) scoring system is an imaging tool that can help distinguish non-muscle-invasive from muscle-invasive disease prior to transurethral resection (TURB). The VI-RADS consists of a five-point scoring system based on the assessment of tumour size, morphology, growth, degree of restriction and contrast capture to assess the likelihood of bladder wall invasion. VI-RADS was an observational, prospective, multicenter, no profit study. The aims of the study was to clarify the clinical validity of the Vesical Imaging-Reporting and Data System (VI-RADS) for the assessment of muscle invasion (MI) status in comparison with transurethral resection of bladder cancer (TURB) and to evaluate the diagnostic accuracy of the score according to the specific tumour location.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected primary bladder cancer at cystoscopy

Exclusion Criteria:

* Impaired renal function
* claustrophobia
* allergy to paramagnetic contrast agent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected primary bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Vescical Imaging-Reporting and Data System (VI-RADS) in predicting muscle-invasive bladder cancer after transurethral resection | up to 12 weeks
  The sensitivity of Vescical Imaging-Reporting and Data System (VI-RADS) in muscle invasion will be evaluated by comparing the score of VI-RADS with the results of biopsy after transurethral resection of bladder cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cecchini, MD, Principal Investigator — IRCCS INRCA, Ancona, Italy
Locations (3):
- Italy (3):
  - AOU Hospital, Ancona
  - IRCCS INRCA Hospital, Ancona
  - Carlo Urbani Hospital, Iesi

IPD SHARING:
Plan to Share IPD: No